CLINICAL TRIAL: NCT06266312
Title: FeAsibility of a PReoperative, Multimodal Lifestyle InterventiOn in Patients With Breast Cancer ReceivIng Neoadjuvant Chemotherapy
Brief Title: Feasibility of a Preoperative, Multimodal Lifestyle Intervention in Patients With Breastcancer
Acronym: APRIORI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nationaal Fonds tegen Kanker (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Maastricht UMC+
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Prehabilitation; Multimodal lifestyle intervention; Preoperative period; Feasibility study; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, single-centre, longitudinal mixed-methods feasibility study will be performed to investigate the feasibility of a multimodal prehabilitation programme consisting of MIET during neoadjuvant intravenous chemotherapy infusion, HITT and strength training during the last six weeks prior to surgery, and optimising nutritional intake throughout the total preoperative period in patients with breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- multimodal lifestyle intervention (Experimental): A group receiving a multimodal prehabilitation programme consisting of three modalities:
  1. MIET during neoadjuvant intravenous chemotherapy infusion
  2. HITT and strength training during the last six weeks prior to surgery
  3. Optimising nutritional intake throughout the total preoperative period
  Interventions: Behavioral: A multimodal prehabilitation programme

INTERVENTIONS:
Behavioral: A multimodal prehabilitation programme — 1. During the weekly chemotherapy infusion (week 10-20), a supervised moderate-intensity endurance training (MIET) on a cycle ergometer is performed (11x):
     * 5 min. warm-up
     * 35 min. cycling at 40-60% of (HR reserve + resting HR)
     * 5-10 min. cool-down
  2. + strength training
  During week 17-22 a supervised high-intensity interval training + strength training programme is performed (8x):
  HITT:
  * 3 min warm-up (20W)
  * 14 intervals (30sec. work intervals at 60% of WRpeak alternates with 60-sec. rest intervals at 20W) --1 min. cool-down
  Muscle strength:
  4 exercises (leg press, chest press, abdominal crunch, lateral pulldown), 3 sets, 8-12 repetitions at 60% of 1-RM.
  3) During 4 consultations with a dietician (week 9, 15, 20, 22) nutritional intake is evaluated and advice is given on energy and protein requirements. Patients are advised to use a digital food diary to record their intake for ≥3 days a week.
  Other Names: Not appliccable

SUMMARY:
The primary objective of this study is to investigate the feasibility of a multimodal prehabilitation programme consisting of MIET during neoadjuvant intravenous chemotherapy infusion, HITT and strength training during the last six weeks prior to surgery, and optimising nutritional intake throughout the total preoperative period in patients with breast cancer with respect to recruitment, adherence, dropout, safety and acceptance. The secondary objective is to provide a preliminary evaluation of participant responses to a preoperative multimodal lifestyle intervention, on cardiorespiratory fitness, muscle strength, nutritional status, and fatigue in patients with breast cancer receiving neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Rationale: Breast cancer is the most common type of cancer among women. The disease and treatment are associated with an increased risk of deterioration in physical fitness, muscle strength, nutritional status (sarcopenic obesity), mental well-being, health-related quality of life (HRQoL) and fatigue. To improve health outcomes, modifiable factors should be intervened as early as possible. The preoperative period during which patients receive neoadjuvant chemotherapy seems ideal to offer a multimodal lifestyle intervention, but is currently hardly used for this purpose. Nutritional status can be optimised through guidance from a dietician and self-monitoring of nutritional intake via a digital food diary. Additionally, offering a moderate-intensity endurance training (MIET) exercise programme during neoadjuvant intravenous chemotherapy infusion enables supervised exercise at a time when patients would otherwise be inactive. It may also improve tumour perfusion, thereby increasing the effectiveness of cytostatic uptake into the tumour and counteracting resistance to cytostatic drugs. The last six weeks prior to surgery can be used to further optimise cardiorespiratory fitness and muscle strength through a high-intensity interval training (HIIT) and strength training programme. Before the effect of a preoperative, multimodal lifestyle intervention in breast cancer patients receiving neoadjuvant chemotherapy can be investigated, its feasibility needs to be investigated first.

Objective: The primary objective of this study is to investigate the feasibility of a multimodal prehabilitation programme consisting of MIET during neoadjuvant intravenous chemotherapy infusion, HITT and strength training during the last six weeks prior to surgery, and optimising nutritional intake throughout the total preoperative period in patients with breast cancer with respect to recruitment, adherence, dropout, safety and acceptance. The secondary objective is to provide a preliminary evaluation of participant responses to a preoperative multimodal lifestyle intervention, on cardiorespiratory fitness, muscle strength, nutritional status, and fatigue in patients with breast cancer receiving neoadjuvant chemotherapy.

Study design: A prospective, single-centre, longitudinal mixed-methods feasibility study.

Study population: Patients with breast cancer scheduled for neoadjuvant chemotherapy and surgery at the MUMC+ Comprehensive Cancer Center.

Intervention: The multimodal lifestyle intervention consists of three modalities. Patients are asked to complete 11 sessions of MIET during intravenous chemotherapy infusion, 8 sessions of HIIT and strength training in the last six weeks prior to surgery, and 4 consultations with a dietician throughout the preoperative period. The MIET training sessions consist of 45-50 minutes training programme on a cycle ergometer during the chemotherapy infusion. The physiotherapist will additionally advise patients to adhere (or build up to) the Nederlandse Norm Gezond Bewegen (NNGB) on remaining weekdays. The HIIT and strength training sessions consist of a 25 minutes training programme performed on a cycle ergometer, followed by four muscle-strengthening exercises. During the consultations with the dietician, patients' energy and protein intake are evaluated and advice is given on how to achieve the calculated energy and protein requirements. To improve patient self-management and empowerment, patients are also advised to use a free digital food diary.

Main study parameters/endpoints: The primary endpoint of the study is the feasibility of the multimodal lifestyle intervention with respect to recruitment, adherence, drop-out, safety and acceptance.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks of participating in the multimodal lifestyle intervention are considered minimal. The performance tests (Steep Ramp Test, 1-Repetition Maximum) are safe and feasible for this population. However, patients could experience some discomfort (exhaustion, muscle fatigue) due to the performance tests or exercise programs. Study related adverse events, related to exercise or nutritional changes, will be closely monitored and managed by the physiotherapist and dietician. Participation in study will take approximately 17.5 to 20 hours per patient. This time includes two consults with a physiotherapist, 8 sessions of HIIT and strength training, 4 consultations with a dietician, filling in the digital food diary and one semi-structured interview with the researcher to investigate acceptance of the multimodal lifestyle intervention and study procedures as perceived by patients. Patients are asked to complete questionnaires on fatigue and nutritional status on five different occasions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage I-III breast cancer eligible for neoadjuvant intravenous chemotherapy at the MUMC+
* Aged ≥18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status Scale grade 0-1 (Table 1)
* Enough understanding of the Dutch language

Exclusion Criteria:

* Human Epidermal growth factor Receptor 2 (HER2) - positive tumour
* Scalp cooling
* Conditions that seriously hamper physical exercise
* Incapacitated subjects as reported by the attending medical specialist in the medical record. When any doubt arises, the patient will not be considered eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate (%) | Week 0
  Number of included patients / number of eligible patients within the study period
Characteristics of included participants | Week 0
  Sex, age, cancer stage, comorbidities (cardiovascular, musculoskeletal, pulmonary, neurological, other).
Attendance rate for MIET sessions (%) | Week 10-20
  Number of attended sessions / total number of planned sessions
Adherence rate, exercise relative dose intensity (ExRDI) MIET (%) | Week 10-20
  ExRDI = completed exercise dose intensity / prescribed exercise dose intensity.
  Completed exercise dose intensity is defined as total duration (min.) performed in targeted HR zones * total training duration (min.) performed.
  Prescribed exercise dose intensity is defined as total duration (min) prescribed in targeted HR zones * prescribed training duration.
  ExRDI MIET = calculated for each participant individually, cumulative for all training sessions; and cumulative for all participants.
Reasons for not having executed a training session as intended | Week 10-20
  Reasons for not having executed a training session as intended (e.g., low saturation, high blood pressure, the intended training intensity could not be sustained, tiredness, etc.)
Attendance rate HIIT + strength sessions (%) | Week 17-22
  Number of attended sessions / total number of planned sessions
Adherence rate, ExRDI HIIT training (%) | Week 17-22
  ExRDI = completed exercise dose intensity / prescribed exercise dose intensity.
  Completed exercise dose intensity is defined as total duration (min) work intervals * completed work rate (W) work interval.
  Prescribed exercise dose intensity is defined as prescribed total duration (min) work intervals * prescribed work rate (W) work interval.
  ExRDI HIIT is calculated for each participant individually, cumulative for all training sessions; and cumulative for all participants.
Adherence rate, ErXDI strength training (%) | Week 17-22
  ExRDI = completed exercise dose intensity / prescribed exercise dose intensity.
  Completed exercise dose intensity is defined as completed training volume (weight * sets * repetitions)
  Prescribed exercise dose intensity is defined as prescribed training volume (weight * sets * repetitions)
  ExRDI strength training is calculated per participant per training session for each exercise and for all four exercises cumulative. And cumulative for all training sessions; and cumulative for all participants.
Attendance rate for dietary consultations (%) | Weeks 9, 15, 20 and 22
  Number of attended sessions / total number of planned sessions
Percentage of use of the digital food diary 'Mijn Eetmeter'(%) | Weeks 15, 20 and 22
  Number of days the food diary is filled out / total number of days agreed to complete
Percentage of days on which nutritional requirements were achieved (%) | Weeks 15, 20 and 22
  Number of days on which individual nutritional recommendations (energy and protein intake) were achieved / number of days on which 'Mijn Eetmeter' is filled out
Reasons for not achieving the nutritional requirements as intended | Weeks 15, 20 and 22
  Reasons for not achieving the nutritional requirement as intended
Drop-out rate (%) | Week 1-22
  Number of participants who dropped out divided by the total number of participants
Time point of drop-out | Week 1-22
  Time point in the study (week number after inclusion) during which patients drop-out
Reasons for drop-out | Week 1-22
  Reasons for drop-out
Serious adverse events (SAE) | Week 10-22
  Any untoward medical occurrence or effect that:
  * results in death;
  * is life threatening (at the time of the event);
  * requires hospitalisation or prolongation of existing inpatients' hospitalisation;
  * results in persistent or significant disability or incapacity;
  * is a congenital anomaly or birth defect; or
  * any other important medical event that did not result in any of the outcomes listed above due to medical or surgical intervention but could have been based upon appropriate judgement by the investigator. An elective hospital admission will not be considered as a serious adverse event.
Study related adverse events | Week 10-22
  Any occurrence of the following study related adverse events during or immediately after a MIET or HITT and strength training session:
  * Early termination of the training, because of the occurrence of one of the subjective or objective termination criteria (as described in section 5.1)
  * extravasation (unintentional leakage of the chemotherapy agent from the vein into the surrounding tissue
  * collapse
  * severe muscle pain lasting >2 days
  * dizziness
  * severe nausea
  * excessive sweating
  * palpitations or chest pain during exertion
Acceptance - Experiences with the multimodal lifestyle intervention | Week 22
  Experiences with the multimodal lifestyle intervention as perceived by patients. Experiences are explored by the researcher through conducting a semi-structured interviews with every patient. Semi-structured, individual, in-depth interviews are conducted in Dutch . Interviews are aimed to last 30 minutes sand will be conducted in a private room at the Department of Physiotherapy of the MUMC+.
  Topic guide:
  * What was your experience with the multimodal lifestyle intervention in general?
  * What was your experience with the Moderate-intensity endurance training (MIET) during intravenous chemotherapy infusion?
  * What was your experience with the High-intensity interval training (HIIT) and strength training
  * What was your experience with the nutritional counselling and use of the digital food diary 'Mijn Eetmeter'?
Acceptance - Suitability of the multimodal lifestyle intervention and study procedures | Week 22
  Suitability of the intervention and study procedures as perceived by patients Suitability is explored by the researcher through conducting a semi-structured interviews with every patient. Semi-structured, individual, in-depth interviews are conducted in Dutch . Interviews are aimed to last 30 minutes sand will be conducted in a private room at the Department of Physiotherapy of the MUMC+.
  Topic guide:
  * Did you consider the intervention to be suitable for patients with breast cancer receiving neoadjuvant chemotherapy?
  * Did you consider the study procedures to be suitable for patients with breast cancer receiving neoadjuvant chemotherapy?
Acceptance - Barriers and enablers regarding participation in the study | Week 22
  Barriers and enablers regarding participation in the study as perceived by patients.
  Barriers and enablers are explored by the researcher through conducting a semi-structured interviews with every patient. Semi-structured, individual, in-depth interviews are conducted in Dutch . Interviews are aimed to last 30 minutes sand will be conducted in a private room at the Department of Physiotherapy of the MUMC+.
  Topic guide:
  * Which factors have positively influenced participation in the intervention?
  * Which factors have negatively influenced participation in the intervention?

SECONDARY OUTCOMES:
Fatigue | Week 0, 9, 17, 20, 22
  Fatique as determined on the Multidimensional Fatigue Index (MFI-20)
Cardiorespiratory fitness | Week 0, 9, 17, 20, 22
  Peak Work Rate (WRpeak) (W/kg) as determined on the Modified Steep Ramp Test (SRT)
Muscle strength | Week 0, 9, 17, 20, 22
  1-repetition maximum (1-RM) (kg) as determined by the Indirect RM tests on the leg press, chest press, abdominal crunch and lateral pulldown strength equipment
Nutritional status | Week 0, 9, 15, 20, 22
  Nutritional status as determined by the Patient Generated Subjective Global Assessment (PG-SGA) short form. The PG-SGA short form results in a PG-SGA score between 0 and 36 with a higher score indicating a higher risk of malnutrition and a higher need to intervene regarding the nutritional status.
  Scoring:
  0-1 = no intervention needed at this time. Regular reassessment during treatment.
  2-3 = education to patient and family by dietitian, nurse, or other healthcare provider with medication intervention as indicated by present symptoms (section 3) and laboratory tests if applicable.
  4-8 = (multidisciplinary) nutritional intervention by dietitian necessary, in combination with nurse or physician as indicated by present symptoms.
  ≥9 = severe indication for improved symptom control and/or nutritional intervention.
Weight (kg) | Week 9, 15, 20, 22
  Weight measured in kg on a weighing scale
Height (cm) | Week 9
  Height measured in centimeters on a stadometer
Body Mass Index (BMI) | Week 9, 15, 20, 22
  Weight / (height*height)
Energy and protein intake (absolute kcal and gr and gr/kg body weight per day) | Week 9, 15, 20, 22
  Determined by self-reported nutritional intake using the 'Mijn Eetmeter' digital food diary on at least three days per week (two weekdays and 1 weekend day)
Energy requirements (kcal) | Week 9
  Calculated using the WHO-formula in patients with a BMI ≤ 30 kg/m2, and using the Harris & Benedict formula in patients with a BMI > 30 kg/m2
Protein requirements | Week 9
  1.2 - 1.5 g protein/ kg body weight per day BMI < 20 kg/m2: calculation based on weight matching a BMI of 20 kg/m2 BMI 20 - 25 kg/m2: calculation based on actual weight BMI > 25 kg/m2: calculation based on fat free mass determined by the formula of Gallagher
Circumference of upper arm and waist (cm) | Week 9, 15, 20, 22
  Circumference of upper arm and waist (cm) measured in stance using a tape measure.

OTHER OUTCOMES:
Chemotherapy Relative Dose Intensity (RDI) | Week 22
  RDI quantifies the total amount of chemotherapy drugs a patient receives relative to the planned or standard dose for a specific treatment regimen. It is calculated by dividing the total actual dose intensity (the total amount of drug received) by the total planned or standard dose intensity (the total intended or recommended amount of drug) * 100. This approach considers the cumulative impact of all chemotherapy sessions and provides a more accurate reflection of the patient's overall exposure to the chemotherapy drugs over the course of treatment.
Treatment-related Side effects | Week 10-22
  Treatment-related side-effects are monitored weekly by the physiotherapist throughout the study period though patient-report.
  * Nausea
  * Vomiting
  * Oral mucositis (painful mouth)
  * Diarrhea
  * Constipation
  * Fever
  * Neutropenic fever
  * Febrile neutropenia
  * Periferal Sensoric neuropathy
  * Handfoot syndrome
  * Fatique
  * Hair loss

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Dijk - Huisman, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
We do not intent to make IPD available to other researchers.